CLINICAL TRIAL: NCT06138418
Title: Spasticity Multidisciplinary Management : QoL and Physical Activity Measurement with Connected Health Devices (PEPS)
Acronym: PEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01629-34
Record Dates: First submitted 2023-07-05; First posted 2023-11-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Spastic Foot
Keywords: spasticity; spastic foot; podometer; neurosurgery
MeSH Terms: conditions — Muscle Spasticity | interventions — Denervation; Tenotomy

STUDY DESIGN:
Intervention Model Description: Longitudinal evaluation waking ability within activity devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Longitudinal cohort study (Experimental): Longitudinal cohort study
  Interventions: Procedure: Neurotomy

INTERVENTIONS:
Procedure: Neurotomy — Surgical treatment of spastic foot
  Other Names: Tenotomy

SUMMARY:
PEPS is a 18 months prospective bicentric study on 30 patients with spastic foot. The main objective is to evaluate the mean daily gait perimeter modifications mesured by connected watch, 6 months after spastic equinus foot surgery versus before this surgery. Investigator will lend a connected watch during the first consultation, and the patient will use it during 10 days in order to collect his mean daily gait perimeter. A lot of other tests will be realised in order to caracterize the clinical picture of each patient. After patients will be operated and all caracteristics of the surgery will be collected. Finally, at 6 months appointment, investigator will do the same analysis than first appointment in order to comparate the data for functional prognosis.

DETAILED DESCRIPTION:
The study is proposed to eligible patients after a pluridisciplinar specialised appointment in the Neurosurgery ward, realised by a neurosurgeon, an orthopedist and a PRM physician. After spastic equinus foot diagnosis needed surgery et after patient's consent to the surgery, investigator will proposed to patient to participate at our study.

Before surgery, demographic datas, spasticity clinical datas, clinical examination (Ashworth and Penn scale), past treatments are collected. Other investigations are realised : FIM, NFAC, Rivermead mobility index, Lower extremity functional scale, SF36, EQ5D. Gait perimeter are collected by the connected watch, and also with a 10 meters test, the gait perimeter on flat and level ground which is unencumbered by any obstacles, Gaitrite evaluation. Patient will conserved the connected watch during all the study duration.

Peroperative datas are collected for each pateints with 3 times. First, before surgery, investigator collect joint range of motion under general anesthesia but without curarization. Second, during surgery, the surgical technique is described, with which nerves and which muscles are treated. Finally, after surgery, investigator will de novo collect joint ranges with the same clinical conditions.

At 6 months appointment, routine datas are collected (surgical complications, clinical examination) and also the notified investifations (FIM, NFAC ...), clinical investigations (Gaitrite, connected watch datas ...)

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Walking patient
* Spastic foot surgery indication
* Consent form ok
* Patient with iOS or Android mobile phone

Exclusion Criteria:

* Previous spastic surgery
* Psychiatric disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Walking perimeter changes measured by a connected watch before vs after spastic foot surgery | 18 months
  Evaluate daily walking perimeter measure measured during 10 days with a connected watch in operated patients between 6 months appointment and pre surgical appointment. Use of appariated Student t test and Spearman test

SECONDARY OUTCOMES:
Diagnostic performance of walking perimeter measure | 18 months
  Spearman test to evaluate diagnostic performance of connected watch datas with clinical datas (Gaitrite, 10 m test ...)
Quality of measure | 18 months
  descriptives statistics on percentage of days when connected watch used
Quality of measure | 18 months
  descriptives statistics on percentage of loss of watch
Quality of measure | 18 months
  descriptives statistics on evaluation of acceptability of connected watch.
Walking perimeter improvement delay after plaster cast remove | 18 months
  daily mean after plaster cast remove in which walking perimeter is increasing for 50%
SF-36 Quality of life evolution before vs after surgery | 18 months
  Student t test to evaluate the QOL modications
EQ5D Quality of life evolution before vs after surgery | 18 months
  Student t test to evaluate the QOL modications
Rivermead Quality of life evolution before vs after surgery | 18 months
  Student t test to evaluate the QOL modications
LEFS Quality of life evolution before vs after surgery | 18 months
  Student t test to evaluate the QOL modications

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel Lemée, MD PHD, Principal Investigator — University Hospital, Angers
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheean G. The pathophysiology of spasticity. Eur J Neurol. 2002 May;9 Suppl 1:3-9; dicussion 53-61. doi: 10.1046/j.1468-1331.2002.0090s1003.x. PMID 11918643
- [Background] Wallace D, Duncan PW, Lai SM. Comparison of the responsiveness of the Barthel Index and the motor component of the Functional Independence Measure in stroke: the impact of using different methods for measuring responsiveness. J Clin Epidemiol. 2002 Sep;55(9):922-8. doi: 10.1016/s0895-4356(02)00410-9. PMID 12393081
- [Background] Milligan J, Ryan K, Lee J. Demythifier la spasticite en premiere ligne. Can Fam Physician. 2019 Oct;65(10):e422-e428. French. PMID 31604751
- [Background] Nikamp CD, Buurke JH, van der Palen J, Hermens HJ, Rietman JS. Early or delayed provision of an ankle-foot orthosis in patients with acute and subacute stroke: a randomized controlled trial. Clin Rehabil. 2017 Jun;31(6):798-808. doi: 10.1177/0269215516658337. Epub 2016 Jul 7. PMID 27390153
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Trompetto C, Marinelli L, Mori L, Pelosin E, Curra A, Molfetta L, Abbruzzese G. Pathophysiology of spasticity: implications for neurorehabilitation. Biomed Res Int. 2014;2014:354906. doi: 10.1155/2014/354906. Epub 2014 Oct 30. PMID 25530960
- [Background] Sankaranarayan H, Gupta A, Khanna M, Taly AB, Thennarasu K. Role of ankle foot orthosis in improving locomotion and functional recovery in patients with stroke: A prospective rehabilitation study. J Neurosci Rural Pract. 2016 Oct-Dec;7(4):544-549. doi: 10.4103/0976-3147.185507. PMID 27695234
- [Background] Deltombe T, Gustin T. Selective tibial neurotomy in the treatment of spastic equinovarus foot in hemiplegic patients: a 2-year longitudinal follow-up of 30 cases. Arch Phys Med Rehabil. 2010 Jul;91(7):1025-30. doi: 10.1016/j.apmr.2010.04.010. PMID 20599040
- [Background] King BW, Ruta DJ, Irwin TA. Spastic foot and ankle deformities: evaluation and treatment. Foot Ankle Clin. 2014 Mar;19(1):97-111. doi: 10.1016/j.fcl.2013.10.007. PMID 24548513
- [Background] Kidd D, Stewart G, Baldry J, Johnson J, Rossiter D, Petruckevitch A, Thompson AJ. The Functional Independence Measure: a comparative validity and reliability study. Disabil Rehabil. 1995 Jan;17(1):10-4. doi: 10.3109/09638289509166622. PMID 7858276
- [Background] Dones I, Nazzi V, Broggi G. The guidelines for the diagnosis and treatment of spasticity. J Neurosurg Sci. 2006 Dec;50(4):101-5. PMID 17108887
- [Background] Menz HB, Latt MD, Tiedemann A, Mun San Kwan M, Lord SR. Reliability of the GAITRite walkway system for the quantification of temporo-spatial parameters of gait in young and older people. Gait Posture. 2004 Aug;20(1):20-5. doi: 10.1016/S0966-6362(03)00068-7. PMID 15196515
- [Background] Rossier P, Wade DT. Validity and reliability comparison of 4 mobility measures in patients presenting with neurologic impairment. Arch Phys Med Rehabil. 2001 Jan;82(1):9-13. doi: 10.1053/apmr.2001.9396. PMID 11239279
- [Background] Rene F, Casimiro L, Tremblay M, Brosseau L, Lefebvre A, Beaudouin M, Belliveau V, Bergeron LP. Une version canadienne francaise du Lower Extremity Functional Scale (LEFS) : L'Echelle fonctionnelle des membres inferieurs (EFMI), partie I. Physiother Can. 2011 Spring;63(2):242-8. doi: 10.3138/ptc.2010-11F. Epub 2011 Apr 13. French. PMID 22379265
- [Background] Ferguson T, Rowlands AV, Olds T, Maher C. The validity of consumer-level, activity monitors in healthy adults worn in free-living conditions: a cross-sectional study. Int J Behav Nutr Phys Act. 2015 Mar 27;12:42. doi: 10.1186/s12966-015-0201-9. PMID 25890168
- [Background] Collen FM, Wade DT, Robb GF, Bradshaw CM. The Rivermead Mobility Index: a further development of the Rivermead Motor Assessment. Int Disabil Stud. 1991 Apr-Jun;13(2):50-4. doi: 10.3109/03790799109166684. PMID 1836787